CLINICAL TRIAL: NCT00654186
Title: A Phase II Study Evaluating the Toxicity and Efficacy of Single Agent Lenalidomide (Revlimid®) in Chemotherapy-Naïve Androgen-Independent Prostate Cancer Patients
Brief Title: Study Evaluating Toxicity & Efficacy of Lenalidomide(Revlimid®)in Chemotherapy-Naïve AIPC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RV-PCA-PI-327
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-02

CONDITIONS: Prostate Cancer
Keywords: Androgen Independent Prostate Cancer (AIPC); Chemo naive
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — 25mg daily on days 1 - 21 followed by 7 days of rest repeated every 28 days
  Other Names: Lenalidomide

SUMMARY:
This is a single institution, open label, phase II study in androgen-independent prostate cancer patients who are chemotherapy-naïve. Patients will receive Revlimid® 25 mg daily on Days 1-21 followed by 7 days of rest repeated every 28 days. Treatment continues until disease progression, patient's withdrawal, unacceptable toxicity or the investigator's discretion.

DETAILED DESCRIPTION:
The standard of care in patients with androgen independent prostate cancer (AIPC) is debated. Systemic chemotherapy has shown a survival advantage with a Taxotere-based regimen, but this therapeutic approach is associated with significant toxicity and morbidity. Furthermore, some patients with AIPC are asymptomatic with minimal disease burden making systemic chemotherapy a less attractive option. Identifying active agents that are effective in this patient population is of vital importance, as this may delay the need to chemotherapy, palliate symptoms, delay progression, and potentially prolong survival. Acceptable approaches in this setting include vaccine therapies, targeted agents, immunotherapy, or non-taxotere based chemotherapeutic programs. Targeted therapy is of particular interest as this usually avoids side effects of chemotherapy by attacking tumor cells and sparing normal tissue. Ongoing research continues to identify pathways by which the prostate cancer cells become refractory to androgen blockade. During the development of prostate cancer, cell survival depends primarily on the androgen receptor, which is bound to heat shock proteins in the cytoplasm. The active metabolite of testosterone, namely dihydrotestosterone (DHT) binds to the receptor relocating it to the nucleus where it dimerizes, activating transcription genes that are involved in the growth and survival of the cancer cell. Plausible etiologies for the development of hormone resistance and continued cell growth despite adequate castration include changes in antigen receptor expression, changes in the receptor structure, and changes in androgen receptor function with more than one mechanism contributing to this resistance. Several investigators have shown that the androgen receptor gene is the only gene that is consistently up regulated during tumor progression. This increase in androgen receptor mRNA and protein was both necessary and sufficient to convert prostate cancer growth from hormone-sensitive to hormone-refractory, and was dependent on a functional ligand-binding domain. Consequently, one can divide mechanisms of androgen resistance into those that involve the androgen receptor and those that do not.Pathways involving the androgen receptor allow for prostate cancer progression through amplification or mutations of the receptor, deregulation of growth factors or cytokines, and alteration of activators. Amplification of the androgen receptor gene leads to enhanced activation of that receptor even at lower levels of androgens. In addition, mutations in the receptor gene allow for activation of the receptor by different ligands. Peptide growth factors, such as insulin-like growth factor, keratinocyte growth factor, epidermal growth factor, and interleukin-6 (IL 6) can activate the antigen receptor independent of androgens.Deregulation of the apoptotic genes is another important pathway in AIPC development. PTEN tumor suppressor gene (Phosphatase and Tensin Homologue) is mutated in AIPC allowing for the loss of the inhibitory effect that it usually exhibits on the phosphatidylinositol 3-kinase pathway, causing overproduction of akt allowing for cell survival to continue. Another deregulated proapoptotic oncogene, namely bcl-2 allows for cell survival and eventually progression of disease. It has been postulated for years that tumors need an alternative source of nutrients once they outgrow their own supply. Folkman suggested that an angiogenic switch takes place, which accelerates tumor proliferation. Inhibiting tumor proangiogenic factors without affecting normal vasculature has become an attractive theory to inhibit tumor growth. Since prostate cancer, like other malignancies, require blood vessel formation to develop metastases, finding methods that would disrupt this process became of paramount importance. Two separate studies have shown that elevated levels of the vascular endothelial growth factor (VEGF) correspond with advanced stage, progression, and poor survival in prostate cancer. Since VEGF is a major regulator of angiogenesis; a process that is increased in AIPC and since VEGF also correlates with increased microvessel density as well as prognosis, a logical step was to evaluate the activity of VEGF inhibitors and other anti-angiogenesis agents in AIPC. Lenalidomide (Revlimid®) is an analogue of thalidomide that has demonstrated enhanced immunomodulatory properties and a more favorable toxicity profile. The fact that AIPC depends on angiogenesis and lack of appropriate immune reaction to malignant cells and the fact that Revlimid® exhibits its activity by inhibiting angiogenesis with appropriate immunomodulation, makes this agent an attractive option to study in this disease setting.Several investigations suggested activity with thalidomide in AIPC but most studies were in patients who have failed systemic chemotherapy. In addition, Revlimid® has been shown in phase I trials to be safe, less toxic and more tolerable than Thalidomide, with potential activity. This study aims at evaluating the toxicity and efficacy of Revlimid® in AIPC patients who are chemotherapy-naive.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form.
2. Age 18 years at the time of signing the informed consent form.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Documented prostate cancer regardless of Gleason score
5. Patients should be considered hormone refractory and androgen independent. They must fail LHRH analogues, and anti-androgen withdrawal trial. Failure is confirmed by an increase in PSA value of 10% or more than the value immediately before, and confirmed by another assessment 2 weeks later that shows a further increase.
6. Patients must have measurable disease either biochemically (using PSA) and/or using the RECIST criteria for visceral organ involvement and/or bone disease
7. ECOG Performance Status of 2 or less.
8. Adequate liver function tests with ALT/AST being < 3x normal, total bilirubin of 1.5 or less, and adequate renal function measured by a creatinine of 2.0 mg/dl or less. Alkaline phosphatase values are never exclusion criteria if it is deemed related to bone metastases.
9. Patients need to have adequate bone marrow function.

   * ANC of 1000 or above,
   * Hgb of 9.0 g/dl or above,
   * Platelets of 100,000 or above. If other causes are affecting plts counts such as autoimmune disorders, patients are allowed on study. Patients with inadequate bone marrow function that is deemed related to bone marrow involvement with prostate cancer are allowed at the investigator's discretion.
10. Patients with other malignancies are allowed as long as there is no evidence of the other malignancy present at entry time, and it has been 3 years or more since the treatment for the other disorder was completed.
11. Patients with prior exposure to investigational therapies including vaccines are allowed on this study as long as their last exposure was 4 weeks prior to study entry. Erlotinib exposure and GM-CSF is not an exclusion criteria as it is not considered chemotherapy.
12. Patients with known bone metastases are allowed to receive intravenous bisphosphonates such as aredia or zometa. Patients on oral bisphosphonates are also allowed.
13. All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®.
14. Patients must agree to use a latex condom during sexual contact with a female of childbearing potential, even if they have had a successful vasectomy. See Appendix: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
15. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).

Exclusion Criteria:

1. Prior systemic chemotherapy for AIPC. Investigational therapy such as vaccines, immunotherapy, and oral targeted agents such as erlotinib, sorafenib, or sunitinib are allowed.
2. Prior exposure to lenalidomide
3. Known HIV positive status
4. Known brain metastases.
5. Steroids are allowed concomitantly ONLY IF they are taken for another chronic medical condition (Such as COPD, Multiple sclerosis…etc)
6. Presence of other malignancies, unless the last treatment received for any other malignancy was 3 years or more. Non-melanoma skin cancers are excluded.
7. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
8. Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study or confounds the ability to interpret data from the study.
9. Use of any other experimental drug or therapy within 28 days of baseline.
10. Known hypersensitivity to thalidomide.
11. Known positive for HIV or infectious hepatitis, type A, B or C

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists, SC
Locations (2):
- United States (2):
  - Oncology Specialists, S.C, Niles, Illinois
  - Oncology Specialists, S.C, Park Ridge, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- Revlimid Oral for 21days: Revlimid: 25mg by mouth daily on days 1 - 21 followed by 7 days of rest repeated every 28 days
Period: Overall Study
Arm/Group | Revlimid Oral for 21days
Started | 32
Completed | 27
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: 32 patients started the study. 27 patients had two or mor cycles of study medication. 5 patients withdrew from the study before completing one cycle, making them not evaluable for response
Arm/Group | Revlimid Oral for 21days
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Clinical Benefit (OCB), Defined as the Sum of Complete Response (CR), Partial Response (PR), and Stable Disease (SD) Divided by the Number of Participants
Description: The OCB was assessed using Recist 1.0 as defined in the protocol. A CR was defined as the disappearance of all lesions. A PR was defined as > or equal to a 30% decrease in the sum of the longest diameter of measureable lesions, SD was defined < a 30% decrease in the sum of the longest diameter of measureable lesions and < a 20% increase in the sum of the longest diameter of measureable lesions. For a CR, PR or SD, there are no new lesions.
  Prostate-Specific Antigen (PSA) was also evaluated. A PSA CR was a PSA < or equal to 4 ng/dl. A PSA PR was a PSA that decreased by > or equal to 50%. Stable PSA was defined as a PSA that increased >25% and decreased < 50%.
Time Frame: 24 months for acrual
Population: evaluable patients
Measure: Number; unit: percentage of patients
Arm/Group | Revlimid Oral for 21days
Number analyzed (Participants) | 27
percentage of patients | 74

2. Secondary Outcome: Time to PSA Progression
Description: As defined in the protocol PSA progression was an increase of at least 25%
Time Frame: 24 months for acrual
Measure: Median (Full Range); unit: months
Arm/Group | Revlimid Oral for 21days
Number analyzed (Participants) | 27
months | 3 [2 to 11]

3. Secondary Outcome: Time to Disesase Progression as Measured by Radiographic Progression
Description: Progressive disease (PD) was determined, as outlined in the protocol, by using Recist 1.0. PD is defined as greater than or equal to a 20% increase in the sum of all measureable lesions or the apprearance of two new bone lesions or the appearnce of one new soft tissue lesion.
Time Frame: 24 months
Measure: Median (Full Range); unit: months
Arm/Group | Revlimid Oral for 21days
Number analyzed (Participants) | 27
months | 4 [2 to 16]

ADVERSE EVENTS:
Groups:
- Revlimid Orally for 21 Days: Revlimid: 25mg daily on days 1 - 21 followed by 7 days of rest repeated every 28 days
Arm/Group | Revlimid Orally for 21 Days
Serious Adverse Events (participants affected / at risk) | 14/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid Orally for 21 Days (N=32)
syncope (Nervous system disorders) | 2 (2)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
atrial fibrilation (Cardiac disorders) | 2 (2)
sepsis (Infections and infestations) | 1 (1)
pancreatitis (Gastrointestinal disorders) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
kidney stones (Renal and urinary disorders) | 1 (1)
bronchitis (Infections and infestations) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
dehydration (Gastrointestinal disorders) | 4 (4)
weakness (General disorders) | 1 (1)
pancytopenia (General disorders) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
rectal abcess (Gastrointestinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
exacerbation of chronic obstructive pulmonary disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
diverticulitis (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid Orally for 21 Days (N=32)
aspartate aminotransferase increased (Hepatobiliary disorders) | 7
atrial fibrilation (Cardiac disorders) | 2
albumin low (Gastrointestinal disorders) | 20
anemia (Blood and lymphatic system disorders) | 22
anxiety (Psychiatric disorders) | 9
anorexia (Gastrointestinal disorders) | 16
arthalgia (Musculoskeletal and connective tissue disorders) | 7
alanine aminotransferase (Hepatobiliary disorders) | 6
Alkaline phosphatase (Hepatobiliary disorders) | 9
back pain (Musculoskeletal and connective tissue disorders) | 7
bruises easily (Blood and lymphatic system disorders) | 8
bleeds easily (Blood and lymphatic system disorders) | 2
bilirubin increased (Renal and urinary disorders) | 2
bloating (General disorders) | 3
constipation (Gastrointestinal disorders) | 29
creatinine increased (Renal and urinary disorders) | 6
congestive heart failure (Cardiac disorders) | 2
cough (Respiratory, thoracic and mediastinal disorders) | 3
cramps (Musculoskeletal and connective tissue disorders) | 2
chills (General disorders) | 5
diarrhea (Gastrointestinal disorders) | 8
diverticulitis (Gastrointestinal disorders) | 3
depression (Psychiatric disorders) | 10
dizziness (General disorders) | 3
dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 5
dehydration (Gastrointestinal disorders) | 6
eyes dry (Eye disorders) | 3
edema (General disorders) | 7
eyes watery (Eye disorders) | 3
fatigue (General disorders) | 23
gynecomastia (General disorders) | 3
globulin low (General disorders) | 2
hyperkalemia (Metabolism and nutrition disorders) | 4
hypoglycemia (Endocrine disorders) | 2
hyperglycemia (Endocrine disorders) | 13
hypokalemia (Metabolism and nutrition disorders) | 7
hematuria (Renal and urinary disorders) | 4
hypotremia (Metabolism and nutrition disorders) | 8
headache (General disorders) | 3
hypocalcemia (Metabolism and nutrition disorders) | 12 (12)
hot flashes (Reproductive system and breast disorders) | 2
hypertension (Cardiac disorders) | 2
hip pain (Musculoskeletal and connective tissue disorders) | 2
itching (Skin and subcutaneous tissue disorders) | 3
insomnia (General disorders) | 5
leukopenia (Blood and lymphatic system disorders) | 18
libido decreased (Reproductive system and breast disorders) | 4
lightheadedness (General disorders) | 5
lymphopenia (Blood and lymphatic system disorders) | 12
leg weakness (General disorders) | 2
mouth dry (Gastrointestinal disorders) | 4
mouth sores (Gastrointestinal disorders) | 2
neutropenia (Blood and lymphatic system disorders) | 18
nausea (Gastrointestinal disorders) | 7
neck sore (Musculoskeletal and connective tissue disorders) | 2
neuropathy motor (Nervous system disorders) | 7
neuropathy sensory (Nervous system disorders) | 3
pain (General disorders) | 5
pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 2
rash (Skin and subcutaneous tissue disorders) | 12
renal insufficiency (Renal and urinary disorders) | 3
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6
syncope (General disorders) | 2
shoulder pain (Musculoskeletal and connective tissue disorders) | 3
skin dry (Skin and subcutaneous tissue disorders) | 6
taste changes (Gastrointestinal disorders) | 6
thrombocytopenia (Blood and lymphatic system disorders) | 20
tachycardia (Cardiac disorders) | 5
throat sore (General disorders) | 3
unrinary tract infection (Infections and infestations) | 3
urinary frequency increased (Renal and urinary disorders) | 3
weight loss (General disorders) | 11
wheezing (Respiratory, thoracic and mediastinal disorders) | 2
weakness (General disorders) | 5
vomiting (Gastrointestinal disorders) | 5
vision problems (Eye disorders) | 2
vision changes (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes